CLINICAL TRIAL: NCT01160510
Title: Genetics of Mammographic Appearances and Patterns (The GenMap Study)
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910137; 10-C-N137
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Benign Breast Disease
Keywords: Breast; Mammographic Density
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Women undergoing mammography: women undergoing mammography at the UVM Breast Cancer Surveillance Consortium site

SUMMARY:
High mammographic density (HMD) is the strongest risk factor for non-familial breast cancer apart from age and gender. Studies of sisters and twins suggest that approximately 67% of the variation in density is attributable to common genetic factors. However, to date, efforts to identify genetic determinants of HMD have achieved limited success. We and others (Boyd et al Lancet Oncol 2009) postulate that this lack of progress in identifying genetic determinants of density is related to a failure to study younger women and misclassification of density. As women age, their breast tissues undergo atrophy, which is manifested radiologically as a decrease in mammographic density, resulting in a convergence of density values and a masking of inter-person variation. This protocol is intended to demonstrate the feasibility of methods that we plan to use in a full-scale analysis of mammographic density among women under age 50 years who receive care at the University of Vermont, Fletcher Allen Health Care (FAHC) and have been followed through the Vermont Breast Cancer Surveillance System (VBCSS).

The Hormonal and Reproductive Epidemiology Branch (HREB) is currently conducting a cross-sectional study entitled, Breast Radiology Evaluation and Study of Tissues (BREAST) Stamp Project which aims to understand why mammographically dense tissues are related to elevated breast cancer risk. This project is being conducted within the VBCSS using breast cancer awareness Stamp Act funds. The BREAST Stamp project has focused on women between the ages of 40-65 years who were referred for radiologically-guided biopsy to evaluate an abnormality identified on a screening mammogram. The study has successfully enrolled over 400 women with collection of questionnaires, buccal and blood samples, and tissues. The study will continue recruiting through May 2010, with a targeted enrollment of 450-500 women. Through the infrastructure developed for the BREAST Stamp Project, mammographic volumetric density data, assessed using a novel method with density phantoms developed at UCSF, has been collected on approximately 25,000 screened women of all ages from February 2008-present.

The current protocol describes a study in which we propose to capitalize on infrastructure that has been established through the BREAST Stamp Project. We propose to perform this study in two phases: Phase one will be a feasibility study: specifically, we propose to demonstrate that we can use a mailing to collect Oragene tube format saliva collection kits as a source of germline DNA and a short self-administered questionnaire. This collection of specimens and data will be used to inform the launch of phase two, the full-scale study to identify determinants of mammographic volumetric density among approximately 10,000 women less than 50 years of age for whom raw images and density data are already collected. During the first phase we hope to demonstrate feasibility by achieving at least 60% participation with unbiased representation of subjects with regard to demographics and volumetric density measurements. Once feasibility of this approach is established, we propose to launch the full-scale study by contacting the remaining (approximately 10,000) women with existing volumetric density data to collect questionnaires and DNA samples necessary to delineate the genetic determinants of mammographic density, as well as to investigate hypothesized risk factors for mammographic density and breast cancer risk, such as alcohol intake, cigarette smoking, and breastfeeding history.

DETAILED DESCRIPTION:
High mammographic density (HMD) is the strongest risk factor for non-familial breast cancer apart from age and gender. Studies of sisters and twins suggest that approximately 67% of the variation in density is attributable to common genetic factors. However, to date, efforts to identify genetic determinants of HMD have achieved limited success. We and others (Boyd et al Lancet Oncol 2009) postulate that this lack of progress in identifying genetic determinants of density is related to a failure to study younger women and misclassification of density. As women age, their breast tissues undergo atrophy, which is manifested radiologically as a decrease in mammographic density, resulting in a convergence of density values and a masking of inter-person variation. This protocol is intended to demonstrate the feasibility of methods that we plan to use in a full-scale analysis of mammographic density among women under age 50 years who receive care at the University of Vermont, Fletcher Allen Health Care (FAHC) and have been followed through the Vermont Breast Cancer Surveillance System (VBCSS).

The study capitalizes on infrastructure that has been established through the BREAST Stamp project that is being carried out in two phases: phase one is a feasibility study: specifically, we propose to demonstrate that we can use a mailing to collect Oragene tube format saliva collection kits as a source of germline DNA and a short self-administered questionnaire. We have completed the phase one feasibility portion of the protocol, which targeted 200 women by mail. As of January 25, 2011, of the 200 that were mailed invitations, 195 women were contacted (5 subjects forms were returned because of bad addresses), and 106 women enrolled. We are currently analyzing data from this feasibility study to determine participation rates, quality of completed questionnaires and saliva samples, and frequencies and distributions of key risk factors and demographics of participants. This collection of specimens and data will be used to inform the launch of phase two, the full-scale study to identify determinants of mammographic volumetric density among 10,000 women less than 50 years of age for whom raw images and density data are already collected.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Women who undergo screening in Vermont are asked about their willingness to participate in research through the VBCSS.
* The phase one feasibility study will enroll women who have agreed to participate in research and were below age 50 years at the time of their screening mammograms between two time periods: February 1, 2008- February 29, 2008 and February 1, 2009- February 28, 2009.

These periods were chosen because all mammograms performed during this interval were performed using Hologic machines equipped with density phantoms as required for this method and these time periods represent the first and second years of density data collection. If the feasibility study proves successful, then phase two of the study will enroll women who have agreed to participate in research and were below age 50 years at the time of their screening mammograms between: February 1, 2008-present time.

EXCLUSION CRITERIA:

-We will exclude women who at the time of their mammogram: had a prior history of breast cancer, had an excisional breast biopsy within the prior year, had implants in place, or had received non-surgical treatments (i.e., systemic therapies or radiation) for cancers of other organs. We will also exclude women who are a participant in the current BREAST Stamp Project.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary clinical (women undergoing mammography at the UVM Breast Cancer Surveillance Consortium site)
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2010-06-24 (Actual); Primary Completion 2012-01-31 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Mammographic density | At Screening
  Mammagraphic density at screening

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Benson, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Vermont Cancer Center - Univ of Vermont, Burlington, Vermont, United States

REFERENCES:
- [Background] Vachon CM, van Gils CH, Sellers TA, Ghosh K, Pruthi S, Brandt KR, Pankratz VS. Mammographic density, breast cancer risk and risk prediction. Breast Cancer Res. 2007;9(6):217. doi: 10.1186/bcr1829. PMID 18190724
- [Background] Kelemen LE, Sellers TA, Vachon CM. Can genes for mammographic density inform cancer aetiology? Nat Rev Cancer. 2008 Oct;8(10):812-23. doi: 10.1038/nrc2466. Epub 2008 Sep 5. PMID 18772892
- [Background] Klifa C, Carballido-Gamio J, Wilmes L, Laprie A, Shepherd J, Gibbs J, Fan B, Noworolski S, Hylton N. Magnetic resonance imaging for secondary assessment of breast density in a high-risk cohort. Magn Reson Imaging. 2010 Jan;28(1):8-15. doi: 10.1016/j.mri.2009.05.040. Epub 2009 Jul 23. PMID 19631485